CLINICAL TRIAL: NCT06735248
Title: A Phase 2, Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study of mRNA-1195 Intramuscular Injection in Participants 18 to ≤55 Years of Age With Multiple Sclerosis
Brief Title: A Study to Investigate Multiple Sclerosis Relapse Prevention With mRNA-1195 Compared With Placebo in Participants Aged 18 to ≤55 Years
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: mRNA-1195-P201; 2024-517949-13-00 (Other: EU CT Number)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; mRNA-1195; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- mRNA-1195 Dose Level 1 (Low Dose) (Experimental): Participants will receive 3 intramuscular (IM) injections at dose level 1 (low dose) on a 0-, 2-, and 6-month schedule.
  Interventions: Biological: mRNA-1195
- mRNA-1195 Dose Level 2 (High Dose) (Experimental): Participants will receive 3 IM injections at dose level 2 (high dose) on a 0-, 2-, and 6-month schedule.
  Interventions: Biological: mRNA-1195
- Placebo (Placebo Comparator): Participants will receive 3 placebo IM injections on a 0-, 2-, and 6-month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1195 — IM injection
  Arms: mRNA-1195 Dose Level 1 (Low Dose); mRNA-1195 Dose Level 2 (High Dose)
Biological: Placebo — IM injection
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate the safety and reactogenicity of mRNA-1195 in participants with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable as determined by Investigator's medical evaluation, which will include assessment of medical history, physical examination, laboratory testing, and review of any previously conducted cardiac monitoring.
* Participants who are Epstein-Barr virus (EBV)-seropositive at screening.
* Participants diagnosed with relapsing multiple sclerosis, including those with a single clinical attack (that is, clinically isolated syndrome [CIS]), as well as participants diagnosed with radiologically isolated syndrome, within 24 months of Screening Visit (that is, early in their multiple sclerosis course) and in the opinion of the Investigator have been neurologically stable for at least 30 days prior to Visit 1/Day 1.
* A participant who could become pregnant is eligible to participate if they are not pregnant or breast/chest feeding and using a highly effective contraceptive method.

Exclusion Criteria:

* Acutely ill or febrile (temperature ≥38.0 degrees Celsius (℃) [100.4 Fahrenheit °F]) within 72 hours prior to or at screening or Day 1.
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* Received or plans to receive any non-study vaccine (including authorized or approved vaccines for the prevention of coronavirus disease 2019 [COVID-19] regardless of vaccine type) within 28 days before or after any study injection, or within 14 days before or after any study injection for the influenza vaccine.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Received systemic immunosuppressants within the 30 day period prior to screening (for corticosteroids, ≥10 milligrams (mg)/day of prednisone or equivalent)
* Participants with any documented history of myocarditis, pericarditis, or myopericarditis.
* Has donated ≥450 milliliter (mL) of blood products within 28 days prior to screening or plans to donate blood products within 28 days post-study injection.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 176 (7 days after each study injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 197 (28 days after each study injection)
Number of Participants with Medically Attended Adverse Events (MAAEs) | Up to Day 347 (up to 6 months after last study injection)
Number of Participants with Adverse Events of Special Interest (AESI), Serious Adverse Events (SAEs) and AEs Leading to Discontinuation of Study Intervention and/or Study Participation | Up to Day 887 (end of study)

SECONDARY OUTCOMES:
Cumulative Number of New Gadolinium (Gd)-enhancing Longitudinal Relaxation Time (T1) Hyperintense Lesions, as Measured by Magnetic Resonance Imaging (MRI) from Baseline to Month 12 and End of Study (Day 887) | Baseline to Month 12 and Day 887 (end of study)
Mean Number of Gd-enhancing T1 Hyperintense Lesions Per Scan, as Measured by MRI from Baseline to Month 12 and End of Study (Day 887) | Baseline to Month 12 and Day 887 (end of study)
Cumulative Number of New and/or Newly Enlarging Transverse Relaxation Time (T2)-weighted Hyperintense Lesions as Measured by MRI from Baseline to Month 12 and End of Study (Day 887) | Baseline to Month 12 and Day 887 (end of study)
Time to First New Disease Activity on Study as Defined by a Clinical Attack Indicative of Central Nervous System (CNS) Involvement at a Site Remote to the First Attack or a New and/or Newly Enlarging T2 or Gd-enhancing Lesion on MRI | Up to Day 887 (end of study)
Geometric Mean Titer (GMT) of B-cell Neutralizing Antibodies (nAbs) and/or Vaccine Antigen-specific Binding Antibodies (bAbs) at Days 1, 85, and 197 | Days 1, 85, and 197
Geometric Mean Fold Rise (GMFR) of B-cell nAbs and/or Vaccine Antigen-specific bAbs at Days 1, 85, and 197 | Days 1, 85, and 197
Change in Expanded Disability Status Scale (EDSS) Score at 3- and 6-month Intervals from Baseline to End of Study (Day 887) | Baseline, Day 887 (end of study)
Time to 6-month Confirmed Disability Progression | Up to Day 887 (end of study)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - Boston Clinical Trials Inc - Internal Medicine, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Sharlin Health & Neurology, Ozark, Missouri
  - Washington University School of Medicine Neurology Clinical Unit, St Louis, Missouri
  - Oklahoma Medical Research Foundation (OMRF) MS Center of Excellence, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - Saturn Research Solutions, Plano, Texas
- University of the Sunshine Coast Clinical Trials, Birtinya, Queensland, Australia
- United Kingdom (8):
  - North Bristol NHS Trust - Southmead Hospital, Bristol
  - Cardiff and Vale University Health Board - University Hospital Wales, Cardiff
  - Anne Rowling Regenerative Neurology Clinic, University of Edinburgh, Edinburgh
  - NHS Greater Glasgow & Clyde - Institute of Neurological Sciences, Glasgow
  - Cambridge Clinical Research Centre, London
  - East Kent Hospitals University NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Sheffield Teaching Hospital NHS foundation Trust, Herries Road, Sheffield